CLINICAL TRIAL: NCT04981041
Title: Escalated Single Platelet Inhibition for One Month Plus Direct Oral Anticoagulation in Patients With Atrial Fibrillation and acUte coRonary Syndrome Undergoing percutaneoUS Coronary Intervention
Brief Title: Escalated Single Platelet Inhibition for One Month Plus NOAC in Patients With Atrial Fibrillation and ACS Undergoing PCI
Acronym: EPIDAURUS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Konstantinos Rizas, PD Dr. med. Konstantinos Rizas, Assistant Professor of Medicine, Co-Principal Investigator, Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EPIDAURUS-2020
Record Dates: First submitted 2021-07-21; First posted 2021-07-28 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Acute Coronary Syndrome; Atrial Fibrillation
MeSH Terms: conditions — Acute Coronary Syndrome; Atrial Fibrillation | interventions — Prasugrel Hydrochloride; Ticagrelor; Clopidogrel

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Potent P2Y12-Inhibition (Experimental): Prasugrel 10mg (5 mg in patients ≥ 75 years old or weighing < 60 kg) q.d. per os or Ticagrelor 90mg bid per os
  Interventions: Drug: Prasugrel or Ticagrelor
- Clopidogrel (Active Comparator): Clopidogrel 75mg q.d. per os
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Prasugrel or Ticagrelor — Escalated antiplatelet therapy with a potent P2Y12- inhibitor for one month in patients with atrial fibrillation and indication for treatment non-vitamin K antagonist oral anticoagulants (NOACs)
  Arms: Potent P2Y12-Inhibition
Drug: Clopidogrel — Clopidogrel and NOAC
  Arms: Clopidogrel

SUMMARY:
The selection of the optimal antithrombotic therapy in patients with nonvalvular atrial fibrillation (AF) and acute coronary syndrome (ACS) undergoing percutaneous coronary intervention (PCI) is challenging. Until recently, triple antithrombotic therapy (TAT) consisting in Aspirin plus Clopidogrel plus OAC was considered the treatment of choice. While efficiently preventing ischaemic events, TAT is associated with an increase in bleeding complications. Therefore, in the past years several randomized controlled trials challenged TAT by comparing a triple antithrombotic therapy (TAT) regimen based on Vitamin K antagonists (VKA) to a dual antithrombotic regimen (DAT) based on non-vitamin K antagonist oral anticoagulants (NOACs) and P2Y12-inhibitors, mainly Clopidogrel in patients with AF undergoing PCI.

However, approximately 30-40% of patients show low response to Clopidogrel and are not adequately protected against ischaemic events, in particular when presenting with ACS. This is supported by a recent meta-analysis reporting that TAT compared to DAT is associated with lower rates of stent thrombosis within 30 days after PCI. It is therefore reasonable to assume that a more potent platelet inhibition within the first month after PCI might reduce the rate of ischaemic complications observed in AF patients undergoing PCI, when receiving DAT. Moreover, a subsequent de-escalation to a less potent platelet inhibition one month after PCI might prevent an increase in bleeding complications.

In EPIDAURUS the investigators will therefore test the hypothesis that DAT using NOAC plus an escalated antiplatelet therapy with a potent P2Y12-inhibitor for one month followed by Clopidogrel reduces ischaemic events without a relevant increase in bleeding complications in patients with AF and ACS undergoing PCI compared to standard DAT with NOAC plus Clopidogrel.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age ≥ 18 years
* Atrial fibrillation requiring oral anticoagulation
* STEMI or NSTEMI (biomarker positive acute coronary syndrome) and successful completion of PCI (randomization will take place within 24h after successful PCI)

Exclusion Criteria:

* Chronic renal insufficiency with glomerular filtration rate < 15 ml/min/1.73m2
* History of ischaemic stroke or transient ischaemic attack (both contraindications for Prasugrel) and history of intracranial bleeding (contraindication for Ticagrelor)
* Contraindication for Clopidogrel or Aspirin
* Contraindication for P2Y12-inhibitor
* Severe chronic liver disease (Child-Pugh C)
* Indication for oral anticoagulation with Vitamin K antagonists
* Moderate to severe mitral stenosis or mechanical heart valve
* Any bleeding BARC type ≥ 2 within the last 4 weeks before index procedure
* Pregnancy or lactation
* Inability to cooperate with the protocol requirements
* Life expectancy < 6 months
* Participation in another investigational drug study
* Previous enrolment in this study
* For women of childbearing potential no negative pregnancy test and no agree to use a reliable method of birth control during the study
* Previous treatment with GP IIb/IIIa inhibitors within the last 12 hours
* A known genetic disorder involved in the metabolism of the study medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2334 (Estimated)
Dates: Start 2021-12-16 (Actual); Primary Completion 2024-12-16 (Estimated); Study Completion 2025-06-16 (Estimated)

PRIMARY OUTCOMES:
Major ischaemic events defined as the composite of all-cause mortality, myocardial infarction, definite or probable stent thrombosis, ischaemic stroke and systemic thromboembolism | 6 weeks
  superiority test
Bleeding type 2 or higher according to the Bleeding Academic Research Consortium (BARC) criteria | 6 weeks
  non-inferiority test

SECONDARY OUTCOMES:
All-cause mortality | 6 weeks
Myocardial infarction | 6 weeks
Definite or probable stent thrombosis | 6 weeks
Ischaemic stroke | 6 weeks
Systemic thromboembolism | 6 weeks
Cardiovascular mortality | 6 weeks
Bleeding type 2 or more according to the Bleeding Academic Research Consortium | 6 weeks
  superiority testing
Urgent revascularization | 6 weeks
All-cause mortality | 6 months
Unplanned hospitalization due to acute heart failure or acute coronary syndrome | 6 months
Ischaemic stroke | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Steffen Massberg, MD, Principal Investigator — LMU Klinikum; Konstantinos Rizas, MD, Principal Investigator — LMU Klinikum
Locations (25):
- Germany (25):
  - Deutsches Herzzentrum München, Munich, Bavaria
  - Universitätsklinikum Freiburg, Universitäts-Herzzentrum Klinik für Kardiologie & Angiologie, Campus Bad Krozingen, Bad Krozingen
  - Kerckhoff-Klinik GmbH, Herzzentrum, Bad Nauheim
  - Campus Benjamin Franklin, Berlin
  - Campus Virchow-Klinikum, Berlin
  - Klinikum Bielefeld gem. GmbH Universitätsklinikum für Kardiologie und Internistische Intensivmedizin, Bielefeld
  - Herzzentrum Dresden GmbH Universitätsklinik an der Technischen Universität Dresden, Klinik für Innere Medizin und Kardiologie, Dresden
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Klinikum Landkreis Erding, Erding
  - Universitätsklinikum Essen, Essen
  - Universitäres Herzzentrum Universitätsklinikum Frankfurt am Main Goethe-Universität, Frankfurt am Main
  - Universitätsklinikum Freiburg, Universitäts-Herzzentrum Klinik für Kardiologie & Angiologie, Campus Freiburg, Freiburg im Breisgau
  - Evangelisches Krankenhaus Hagen-Haspe gGmbH, Klinik für Kardiologie und Rhythmologie, Hagen
  - Medizinische Hochschule Hannover,Zentrum für Innere Medizin, Hanover
  - Universitätsklinikum Heidelberg, Klinik für Kardiologie, Angiologie, Pneumologie, Heidelberg
  - Universitätsklinikum Schleswig-Holstein -Campus Kiel- Klinik für Innere Medizin III mit den Schwerpunkten Kardiologie, Angiologie und internistische Intensivmedizin, Kiel
  - Herzzentrum Leipzig, Universitätsklinik für Kardiologie, Leipzig
  - Universitätsmedizin Mainz, Zentrum für Kardiologie - Kardiologie I, Mainz
  - LMU-Klinikum Campus Grosshadern, Munich
  - LMU-Klinikum Campus Innenstadt, Munich
  - Klinikum Nürnberg Süd, Klinik für Innere Medizin 8, Schwerpunkt Kardiologie, Nuremberg
  - Universitätsmedizin Rostock, Zentrum Innere Medizin, Abteilung Kardiologie, Rostock
  - HBK Hegau-Bodensee Klinikum Singen, Singen
  - Barmherzige Brüder, Klinikum St. Elisabeth Straubing GmbH, II. Medizinische Klinik Innere Medizin, Kardiologie, Intensivmedizin, Pneumologie, Nephrologie und Angiologie, Straubing
  - Universitätsklinikum Tübingen, Tübingen

IPD SHARING:
Plan to Share IPD: No